CLINICAL TRIAL: NCT04591704
Title: The Effect of Diabetes Mellitus on the Morbidity and Mortality Rates in Patients With COVID-19
Brief Title: The Effect of Diabetes Mellitus on the Prognosis of Patients With COVID-19
Acronym: COVID-19-DM2
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Uşak University (Other)
Responsible Party: Sponsor
Other Study IDs: UU-DM003
Record Dates: First submitted 2020-10-16; First posted 2020-10-19 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-05

CONDITIONS: Covid19; Diabetes Mellitus
MeSH Terms: conditions — COVID-19; Diabetes Mellitus | interventions — Hospitalization; Mortality

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Diabetic groups: COVID-19 patients with diabetes mellitus
  Interventions: Other: hospitalisation, necessity of ICU, mortality rate, lung involvement
- Control groups: COVID-19 patients without diabetes mellitus
  Interventions: Other: hospitalisation, necessity of ICU, mortality rate, lung involvement

INTERVENTIONS:
Other: hospitalisation, necessity of ICU, mortality rate, lung involvement — hospitalisation, necessity of ICU, mortality rate, lung involvement

SUMMARY:
All hospitalised patients with COVID-19 who have positive RT-PCR for SARS-COV-2 will be included in the study.

The patients will be divided into two groups, as diabetics and non-diabetics. The COVID-19 patients' medical records will be evaluated and compared in terms of the duration of hospitalization, the presence of lung involvement in Computerised Tomography, the need for intensive care unit and mortality rates in patients with and without diabetes.

DETAILED DESCRIPTION:
All hospitalised patients with COVID-19 who have positive RT-PCR for SARS-COV-2 will be included in the study.

The patients will be divided into two groups, as diabetics and non-diabetics. The diagnosis of diabetes mellitus will be extracted from the medical records and medical history of the patients hospitalised with COVID-19.

The COVID-19 patients medical records will be evaluated and compared in terms of the duration of hospitalization, the presence of lung involvement in Computerised Tomography, the need for intensive care unit and mortality rates in patients with and without diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized for COVID-19

Exclusion Criteria:

* Patients with known malignancy
* Pregnant patients

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients aged between 18-80 years, diagnosed and hospitalised for COVID-19 will be enrolled in to the study
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2020-03-20 (Actual); Primary Completion 2020-10-15 (Actual); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
Duration of Hospitalisation | 1 year
  The time between admission to hospital and discharge
The need for ICU | 1 year
  The admission of hospitalized patients to the intensive care unit.
Mortality | 1 year
  Mortality rates of patients
Lung involvement | 1 year
  The presence of lung involvement on thorax CT

CONTACTS AND LOCATIONS:
Overall Officials: Cevdet Duran, Principal Investigator — Uşak Üniversitesi Tıp fak
Locations (1):
- Usak University Training and Research Hospital, Uşak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No